CLINICAL TRIAL: NCT03627858
Title: A Prospective Non-interventional Study in Patients With Chronic Obstructive Pulmonary Disease That Evolve to Fixed Long-acting Muscarinic Antagonist/Long-acting beta2-agonist/Inhaled Corticosteroid Triple Therapy, Trimbow®
Brief Title: Fixed Dose Triple Therapy in Severe Chronic Obstructive Pulmonary Disease in a Real World Setting
Acronym: TRIVOLVE
Status: Completed | Type: Observational
Sponsor: Chiesi SA/NV (Other)
Responsible Party: Sponsor
Other Study IDs: CHIESI_NIS_0001
Record Dates: First submitted 2018-05-29; First posted 2018-08-14 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: beclomethasone / formoterol / glycopyrronium — As this is a non-interventional study, all treatment decisions will be made at the discretion of the treating physician prior to enrolment in the study and during the entire period of the study. Treatment will be prescribed according to the product label in the summary of product characteristics.
  Other Names: Trimbow®

SUMMARY:
The rationale for this non-interventional study in confirmed moderate to severe chronic obstructive pulmonary disease patients aged 40 years and above, is to assess real-life effectiveness and safety of Trimbow® in clinical practice, and to bridge the gap with the existing clinical data.

DETAILED DESCRIPTION:
This non-interventional study assesses the real-life effectiveness and safety of the fixed triple therapy Trimbow® compared to free triple therapy, considering patient individual data, in clinical practice at second and thirdline centres in patients with confirmed moderate to severe chronic obstructive pulmonary disease.

This is an hypothesis generating study. No formal primary endpoint is defined; parameters are evaluated in an exploratory or descriptive manner.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent
* Patient is aged 40 years or older at time of initiation of Trimbow® treatment
* Patient is diagnosed with moderate or severe chronic obstructive pulmonary disease confirmed by spirometry (post-bronchodilation) based on the Global Initiative for chronic obstructive lung disease (GOLD) 2018 classification
* Patient treated with double inhalation or free triple therapy (using at least 2 devices) who are prescribed Trimbow®

Exclusion Criteria:

• Hypersensitivity to the active substances or to any of the excipients listed below:

* Ethanol anhydrous
* Hydrochloric acid
* Norflurane (propellant)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 40 years or above diagnosed with chronic obstructive pulmonary disease confirmed by spirometry (post-bronchodilation) who were prescribed Trimbow®
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Inhalation technique score | up to 6 months
  Change in Inhalation Technique Score, measured as percentage of correct steps on the Inhalation Checklist (itemized instructions of inhaler correct use per respective Summaries of Product Characteristics) at each routine follow-up visit up to 6 months versus baseline.
  This is an hypothesis generating study. No formal primary endpoint is defined; parameters are evaluated in an exploratory or descriptive manner.

SECONDARY OUTCOMES:
Treatment adherence score | up to 6 months
  Degree of treatment adherence measured via the mean score on the Test of Adherence to Inhalers (TAI) questionnaire, including 5 questions completed by the patient (each item scored from 1 (worst) to 5 (best) with a range from 10 to 50) and 2 items completed by the physician (each item scored 1 (bad) or 2 (good) with a range from 2 to 4) at baseline and each routine follow-up visit up to 6 months versus baseline.
Number of inhaled doses recorded by dose counter since previous visit | up to 6 months
  Number of inhaled doses recorded by dose counter of the inhaler since previous visit, at the first and second routine follow-up visit.
Patient's treatment satisfaction score using visual analogue scale (0-10) | up to 6 months
  The patient's treatment satisfaction score measured on a visual analogue scale from 0 (worst) to 10 (best), at baseline and each routine follow-up visit.
Number of rescue medication used within 7 days prior to each visit | up to 6 months
  The number of rescue medication used within 7 days prior to each visit, recorded at baseline and each routine follow-up visit.
Patient's lung function as measured by spirometry | up to 6 months
  The pre and post bronchodilator forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) are measured at baseline and each routine follow-up visit.
Symptoms score by the Chronic obstructive pulmonary disease Assessment Test (CAT) questionnaire | up to 6 months
  Patients complete the 8-item CAT questionnaire at baseline and each follow-up visit. Total scores range from 0 to 40 and higher scores indicate a worse health status.

OTHER OUTCOMES:
Number of moderate and severe exacerbations at baseline (12 months prior to start) and last follow-up visit | up to 6 months
  The number of moderate and severe exacerbations that occurred within the previous year is collected at the baseline visit and the number of moderate and severe exacerbations occurring during the study is collected at the final visit. Moderate exacerbations are defined as exacerbations that require oral corticosteroid and/or antibiotic treatment. Severe exacerbations are defined as exacerbations that require oral corticosteroid and/or antibiotic treatment plus hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Brusselle, MD-PhD, Principal Investigator — University Ghent
Locations (15):
- Belgium (15):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - GZA Campus Sint-Vincentius, Antwerp
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Clinique Notre-Dame de Grâce ASBL Gosselies, Charleroi
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHR de la Citadelle, Liège
  - AZ Sint-Maarten, Mechelen
  - Hôpital André Vésale, Montigny-le-Tilleul
  - Clinique Saint-Luc Bouge, Namur
  - AZ Delta, Roeselare
  - Hospital Center De Wallonie Picarde, Tournai

IPD SHARING:
Plan to Share IPD: No